CLINICAL TRIAL: NCT00332735
Title: Spinal Anesthesia With 5% Articaine and 0.5% Bupivacaine for Outpatient Lower Limb Surgery. A Double-Blind Randomised Clinical Trial
Brief Title: Spinal Anesthesia With Articaine and Bupivacaine for Outpatient Lower Limb Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reinier de Graaf Groep (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: METC-nr 06-010
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Spinal Anesthesia
Keywords: spinal; anesthesia; articaine; bupivacaine; outpatient; surgery; limbs

INTERVENTIONS:
Drug: spinal administration of articaine
Drug: spinal administration of bupivacaine

SUMMARY:
The purpose of the trial is to compare two local anesthetics, articaine and bupivacaine for outpatient lower limb surgery. Onset and recovery times of sensory and motor blockade will be compared.

DETAILED DESCRIPTION:
The purpose of the trial is to compare two local anesthetics, articaine and bupivacaine for outpatient lower limb surgery.

Faster onset and shorter elimination time favours a short-acting local anaesthetic for spinal anesthesia for out-patient lower limb surgery, e.g. knee arthroscopy, foot and varices surgery. Patients will recover faster and less complications will be expected.

Articaine is said to act faster and shorter than a low dose of bupivacaine. There are not enough data available to establish that articaine is as safe as and more effective by outpatient lower limb surgery than bupivacaine.

Spinal anesthesia with articaine will be compared to spinal anesthesia with bupivacaine in a randomized double blind clinical trial.

Endpoints are:

* onset of sensory and motor block
* maximum spread of sensory level
* recovery from sensory and motor block
* time to micturition
* complications

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Patients planned for an outpatient lower limb surgery
* Procedure under spinal anesthesia
* Informed consent

Exclusion Criteria:

* Contra-indications spinal anesthesia
* History of allergic reactions on amide-type local anesthetics
* Length < 1.60 m or > 1.90 m
* BMI < 18.5 kg/m2 or > 35 kg/m2
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-05; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
recovery time from motor blockade

SECONDARY OUTCOMES:
onset of sensory and motor blockade
maximum spread of sensory blockade (30 min after spinal injection of anesthetic)
spread of sensory blockade after 1,5 hour
recovery time from sensory blockade
time to micturation
complications

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Dijkstra, drs, Principal Investigator — Reinier de Graaf Groep
Locations (1):
- Reinier de Graaf Groep, Voorburg, South Holland, Netherlands

REFERENCES:
- [Background] Vree TB, Gielen MJ. Clinical pharmacology and the use of articaine for local and regional anaesthesia. Best Pract Res Clin Anaesthesiol. 2005 Jun;19(2):293-308. doi: 10.1016/j.bpa.2004.12.006. PMID 15966499
- [Background] Alston RP. Spinal anaesthesia with 0.5% bupivacaine 3 ml: comparison of plain and hyperbaric solutions administered to seated patients. Br J Anaesth. 1988 Oct;61(4):385-9. doi: 10.1093/bja/61.4.385. PMID 3190969
- [Background] Axelsson KH, Widman GB, Sundberg AE, Hallgren S. A double-blind study of motor blockade in the lower limbs. Studies during spinal anaesthesia with hyperbaric and glucose-free 0.5% bupivacaine. Br J Anaesth. 1985 Oct;57(10):960-70. doi: 10.1093/bja/57.10.960. PMID 4041323
- [Background] Kaukinen S, Eerola R, Eerola M, Kaukinen L. A comparison of carticaine and lidocaine in spinal anaesthesia. Ann Clin Res. 1978 Aug;10(4):191-4. PMID 360957